CLINICAL TRIAL: NCT03713229
Title: A Study to Screen for Anal Precancerous Squamous Intraepithelial Lesions and to Prevent Anal Cancer in a Real-life Setting of People Living With HIV at Different Risk: the Seville HIV Anal Cohort
Brief Title: Seville Cohort of People Living With HIV at Risk for Anal Cancer
Acronym: SeVIHanal
Status: Enrolling by invitation | Type: Observational
Sponsor: Hospitales Universitarios Virgen del Rocío (Other)
Collaborators: Instituto de Biomedicina de Sevilla (Unknown)
Responsible Party: Principal Investigator, Karin Neukam, PharmD, PhD, Hospitales Universitarios Virgen del Rocío
Other Study IDs: SeVIHanal Cohort
Record Dates: First submitted 2018-10-18; First posted 2018-10-19 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Anal Squamous Intraepithelial Neoplasia
Keywords: anal squamous intraepithelial lesions; anal squamous cell carcinoma; high-resolution anoscopy; liquid-based cytology; human papillomavirus; men who have sex with men; HIV infection; diagnostic performance
MeSH Terms: conditions — Anus Neoplasms; Homosexuality; HIV Infections | interventions — Mass Screening

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — anal biopsy
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- HIV-infected men who have sex with men: HIV-infected male patients who refer to conducting sexual risk practices that enable HPV transmission
  Interventions: Diagnostic Test: Screening for anal squamous intraepithelial lesions
- HIV-infected men: HIV-infected male patients who neglect conducting sexual risk practices that enable HPV transmission
  Interventions: Diagnostic Test: Screening for anal squamous intraepithelial lesions
- HIV-infected women: HIV-infected female patients disregarding sexual risk practices
  Interventions: Diagnostic Test: Screening for anal squamous intraepithelial lesions

INTERVENTIONS:
Diagnostic Test: Screening for anal squamous intraepithelial lesions — digital-anorectal exam, liquid-based cytology, human papillomavirus testing, high-resolution anoscopy

SUMMARY:
There is increasing awareness of augmenting risk of anal cancer in people living with HIV, especially among men who have sex with men (MSM). High resolution anoscopy (HRA) represents the gold standard to detect pre-cancerous anal high-grade squamous intraepithelial lesions (HSIL), however, the procedure is time-consuming, costly and, most importantly, the learning curve is very flat. This yields a poor implementation of anal screening and, likely, to an excess of otherwise preventable anal cancer. Other screening methods include digital ano-rectal examination, anal-rectal cytology and human papillomavirus (HPV) genotyping, since infection with high-risk HPV genotypes has been identified as the main reason for the development of HSIL. To date, there is no consensus in screening strategies. Furthermore, it remains unclear whether, in whom and to which extend the currently available topic and invasive treatment options for HSIL should be applied, given that the natural history of the development of anal cancer remains poorly understood. The present cohort study aims to provide real-life data on the screening, management and follow-up of HIV-infected MSM is warranted for a better understanding of anal cancer in this setting.

DETAILED DESCRIPTION:
The development of anal precancerous squamous intraepithelial lesions (SIL) and cancer of the anus is mainly caused by infection with high-risk human papillomavirus genotypes (HR-HPV). There is increasing awareness of marked (40 to 130-fold) risk of anal cancer in people living with HIV, especially among men who have sex with men (MSM). With the changing scenario of comorbidities in the HIV-infected population, given the success of modern antiretroviral therapy, anal cancer has emerged as a leading neoplasia across different cohorts in Western countries. In 2014, almost 30000 people were newly diagnosed with HIV in Europe, the majority of cases (77%) being men. This was largely driven by HIV transmission between MSM, which accounted for 42% of all HIV diagnoses. Hence, the incidence of anal cancer is likely to increase in the years to come.

The number of experts who support the necessity of implementing wide programs of anal cancer screening in at-risk populations is rapidly growing. Indeed, both the European Guidelines for treatment of HIV-infected adults and the Guidelines of the Spanish AIDS Society (GESIDA) currently recommend the screening of anal cancer in HIV-infected subjects at risk. It is likely that in years to come, a general recommendation to screen for anal cancer in patients with different conditions associated with immunosuppression is established, as experienced in other populations. In this context, since HIV-negative MSM and women with a history of anogenital dysplasia, as well as transplant patients, exhibit excess risk of anal cancer, these populations have been typically screened in center with ongoing anal cancer screening programs.

Digital ano-rectal examination (DARE) is mainly accepted as the first screening procedure for anal high-risk SIL (HSIL), followed by anal-rectal cytology. Both represent simple methods, however, cytology shows an alarmingly low negative predictive value and furthermore, in case of an abnormal cytology, the patient is referred to high resolution anoscopy (HRA) for biopsy of acetowhite lugol-negative lesions in the anal epithelium, suggestive of HSIL. HRA performance is similar to cervical colposcopy, but unfortunately, the training process is by far longer, hampering its implementation and availability to highly-specialized centers with large cohorts of people living with HIV under care.

Although histological HSIL was identified as precursor of anal cancer, it remains unclear if, which and in whom treatment is indicated, since not all patients progress, a considerable proportion even regresses spontaneously and recurrence rates are high. Treatments currently available include topical imiquimod or 5-fluorouracil, as well as surgical treatment. Due to the lack of data, no consensus of HSIL management has been reached.

Taken together what was mentioned above, real-life data on the screening, management and follow-up of HIV-infected MSM is warranted for a better understanding of anal cancer in this setting.

ELIGIBILITY:
Inclusion Criteria:

* HIV infection as confirmed by ELISA and western blot

Exclusion Criteria:

* Unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV-infected patients seen at the sexually transmitted diseases/HPV consultancy of the Infectious Diseases Unit of the Virgen del Rocío Hospital in Seville, Spain.
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2010-09-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Frequency of anal HSIL | 2007-2025
  The proportion of patients with cancer of the anal squamous intraepithelial cells stage 0, defined as anal high-risk squamous intraepithelial lesions (HSIL) according to the Lower Anogenital Squamous Terminology.
Incidence of anal cancer | 2007-2025
  Incidence rates per person-years of cancer of the anal squamous intraepithelial cells stage 1-4 observed over time as defined by the National Cancer Institute of the National Institutes of Health, US Department of Health and Human Services (www.cancer.gov).

CONTACTS AND LOCATIONS:
Overall Officials: Pompeyo Viciana, MD, PhD, Study Director — Clínica El Sur; Karin Neukam, PharmD, PhD, Study Chair — Hospitales Universitarios Virgen del Rocío; César Sotomayor de la Piedra, Principal Investigator — Hospitales Universitarios Virgen del Rocío
Locations (1):
- Virgen del Rocio University Hospital, Seville, Spain

REFERENCES:
- [Result] Wei F, Gaisa MM, D'Souza G, Xia N, Giuliano AR, Hawes SE, Gao L, Cheng SH, Dona MG, Goldstone SE, Schim van der Loeff MF, Neukam K, Meites E, Poynten IM, Dai J, Combes JD, Wieland U, Burgos J, Wilkin TJ, Hernandez AL, Iribarren Diaz M, Hidalgo-Tenorio C, Valencia Arredondo M, Nyitray AG, Wentzensen N, Chow EP, Smelov V, Nowak RG, Phanuphak N, Woo YL, Choi Y, Hu Y, Schofield AM, Woestenberg PJ, Chikandiwa AT, Hickey AC, de Pokomandy A, Murenzi G, Pere H, Del Pino M, Ortiz AP, Charnot-Katsikas A, Liu X, Chariyalertsak S, Strong C, Ong JJ, Yunihastuti E, Etienney I, Ferre VM, Zou H, Segondy M, Chinyowa S, Alberts CJ, Clifford GM. Epidemiology of anal human papillomavirus infection and high-grade squamous intraepithelial lesions in 29 900 men according to HIV status, sexuality, and age: a collaborative pooled analysis of 64 studies. Lancet HIV. 2021 Sep;8(9):e531-e543. doi: 10.1016/S2352-3018(21)00108-9. Epub 2021 Jul 30. PMID 34339628
- [Result] Milanes Guisado Y, Sotomayor C, Fontillon M, Dominguez Castano A, Espinosa N, Roca C, Lopez-Cortes LF, Viciana P, Neukam K; SeVIHanal Study Group. Incidence Rate and Risk Factors for Anal Squamous Cell Carcinoma in a Cohort of People Living With HIV from 2004 to 2017: Implementation of a Screening Program. Dis Colon Rectum. 2022 Jan 1;65(1):28-39. doi: 10.1097/DCR.0000000000002218. PMID 34694279
- [Result] Viciana P, Milanes-Guisado Y, Fontillon M, Dominguez Castano A, Sotomayor C, Espinosa N, Lopez-Cortes LF, Neukam K. High-risk Human Papilloma Virus Testing Improves Diagnostic Performance to Predict Moderate- to High-grade Anal Intraepithelial Neoplasia in Human Immunodeficiency Virus-infected Men Who Have Sex With Men in Low-to-Absent Cytological Abnormalities. Clin Infect Dis. 2019 Nov 27;69(12):2185-2192. doi: 10.1093/cid/ciz144. PMID 30770528
- [Result] Neukam K, Milanes Guisado Y, Fontillon M, Merino L, Sotomayor C, Espinosa N, Lopez-Cortes LF, Viciana P; SeVIHanal Study Group. High-resolution anoscopy in HIV-infected men: Assessment of the learning curve and factors that improve the performance. Papillomavirus Res. 2019 Jun;7:62-66. doi: 10.1016/j.pvr.2019.01.003. Epub 2019 Feb 1. PMID 30716543